CLINICAL TRIAL: NCT06697080
Title: A Randomized-controlled Clinical Trial to Treat Chinese Advanced AGA With Umbilical Cord-derived Mesenchymal Stem Cell Exosomes
Brief Title: Umbilical Cord-derived Mesenchymal Stem Cell Exosomes on Hair Growth in Patients With Androgenetic Alopecia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: NFEC-2024-323
Record Dates: First submitted 2024-11-17; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Androgenic Alopecia
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Group A visited the clinic once each in the first, second, and third months for treatment with exosomes
  Interventions: Drug: Human umbilical cord mesenchymal stem cells
- Group B (Experimental): Group B visited the clinic twice each in the first, second, and third months for treatment with exosomes.
  Interventions: Drug: Human umbilical cord mesenchymal stem cells

INTERVENTIONS:
Drug: Human umbilical cord mesenchymal stem cells — Human umbilical cord mesenchymal stem cells

SUMMARY:
A total of 50 patients with androgenetic alopecia were selected for the study. Patients who met the inclusion/exclusion criteria were randomly assigned to groups A and B in a 1:1 ratio to receive treatment, with the enrollment date designated as Day 1. Group A visited the clinic once each in the first, second, and third months for treatment with exosomes, while Group B visited the clinic twice each in the first, second, and third months for treatment with exosomes. At the time points of 1, 2, 3, and 6 months after the start of the treatment period, dermatoscopic examinations were conducted on patients in both groups. The differences in hair growth density, hair shaft thickness, and follicle counts within a 1 cm diameter area were compared between the two groups. Additionally, the data differences for each subject at baseline and at the end of the experiment were also assessed.

ELIGIBILITY:
Inclusion Criteria:Clinical diagnosis of Androgenic alopecia · AGA classification include：The No grade for male hair loss was II-V, and the Ludwig grade for female hair loss was I-III Exclusion Criteria: (1) Using medications or supplements, including finasteride, dutasteride, minoxidil or any other hormonal products, that can affect hair growth; · (2) Patients with severe diseases, immune diseases, endocrine diseases and nervous system diseases; (3) Patients with infection, allergic disease and malignant tumor

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2024-06-28 (Actual); Primary Completion 2024-09-28 (Actual); Study Completion 2024-12-28 (Estimated)

PRIMARY OUTCOMES:
hair diameters changed over time | 0 days, 1 month, 3 months, 6 months
  hair diameters changed over time

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Plastic and Aesthetic Surgery, Nanfang Hospital Southern 8 Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No